CLINICAL TRIAL: NCT01150695
Title: A Phase II, Multi-Center, Double-Blind, Randomized Trial Comparing the Safety and Immunogenicity of a Francisella Tularensis Live Vaccine Strain (LVS) Vaccine Produced by DynPort Vaccine Company (DVC-LVS) to a LVS Vaccine in Use by the United States Army Medical Research Institute of Infectious Diseases (USAMRIID-LVS)
Brief Title: Phase II Tularemia Vaccine Comparison
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 08-0006
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2013-03

CONDITIONS: Tularaemia
Keywords: vaccine, Francisella tularensis, Tularemia, rabbit fever, parent protocol
MeSH Terms: conditions — Tularemia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group A (DVC-LVS) (Experimental): Single dose of the Dynport Vaccine Company Live Vaccine Strain (DVC-LVS) product in one arm and normal saline (NS) control in the other arm on Day 0.
  Interventions: Other: Placebo; Biological: Undiluted Francisella tularensis live attenuated vaccine
- Group B (USAMRIID-LVS) (Experimental): Single dose of the United States Army Medical Research Institute of Infectious Diseases Live Vaccine Strain (USAMRIID-LVS) product in one arm and normal saline (NS) control in the other arm on Day 0.
  Interventions: Other: Placebo; Biological: Undiluted Francisella tularensis live attenuated vaccine

INTERVENTIONS:
Other: Placebo — Normal saline will be administered to all subjects as a control and will be given at the same visit as the vaccine (Day 0).
Biological: Undiluted Francisella tularensis live attenuated vaccine — Undiluted Francisella tularensis live attenuated vaccine [approximately 1x10^9 colony forming units (cfu)/mL] produced by Dynport Vaccine Company. Administered by scarification in the ulnar aspect of the volar surface (palm side) of the forearm midway between the wrist and the elbow.
  Arms: Group A (DVC-LVS)
Biological: Undiluted Francisella tularensis live attenuated vaccine — Undiluted Francisella tularensis live attenuated vaccine (approximately 1x10^9 cfu/mL) in use by the United States Army Medical Research Institute of Infectious Diseases. Administered by scarification in the ulnar aspect of the volar surface (palm side) of the forearm midway between the wrist and the elbow.
  Arms: Group B (USAMRIID-LVS)

SUMMARY:
The purpose of this study is to compare 2 experimental vaccines that could provide protection from the disease, tularemia. This research will compare the ability of the vaccines to cause the body to develop an immune (protective) response and obtain more information on side effects of the vaccines. About 220 male and non-pregnant female volunteers 18 to 45 years will participate. Volunteers will be assigned to 1 of 2 vaccine groups by chance. About half of the volunteers will be placed in the DVC-LVS vaccine group and half of volunteers will be placed in the USAMRIID-LVS vaccine group. Additionally, both groups will receive an injection of placebo (inactive salt water). Study procedures include physical exam and blood and urine samples. Evaluation of the vaccination sites will be performed as well as blood samples to measure the body's response to the vaccine. Participants will be involved in the study for about 6 months.

DETAILED DESCRIPTION:
Francisella (F.) tularensis is the organism responsible for tularemia. The organism can infect many different vertebrate and invertebrate hosts, but mostly rodents and lagomorphs. Transmission to humans is generally via an insect vector, such as ticks, mosquitoes, and biting flies, or from handling contaminated animal products or carcasses. F. tularensis is a highly infectious bacterium, with human infection and disease occurring with as few as 10 organisms, and mortality rates approaching 30 percent if untreated. Clinical presentation of tularemia varies in severity depending on the virulence of the organism, the route of entry, the extent of system involvement, and the immune status of the host. Following an incubation period of 3 to 5 days, individuals have an abrupt onset of fever, chills, headache, malaise, anorexia, and fatigue. The clinical presentation of the disease can include one or more the following forms: ulceroglandular (the most common form of the disease), glandular, oculoglandular, pharyngeal, gastrointestinal, pneumonic or typhoidal. This study is a Phase II, multi-center, double-blind, randomized, trial comparing the safety and immunogenicity of a Francisella tularensis live vaccine strain (LVS) vaccine produced by DynPort Vaccine Company (DVC-LVS) to a LVS vaccine in use by the United States Army Medical Research Institute of Infectious Diseases (USAMRIID-LVS). Study Group A will include 110 volunteers who will be vaccinated with a single dose of the DVC LVS product in one arm and normal saline (NS) control in the other arm on Day 0. Group B will include 110 volunteers who will be vaccinated with a single dose of the USAMRIID-LVS product in one arm and normal saline (NS) control in the other arm on Day 0. Both vaccines will be administered by scarification. Approximately 100 microliters aliquot will be withdrawn and placed on the skin, a bifurcated needle will then be used to puncture the skin 15 times through the droplet. The primary objectives are: (Safety): assess the frequency of serious adverse events (SAEs) and Grade 3 and 4 laboratory values following vaccination with either DVC-LVS or USAMRIID-LVS vaccine; (Take): assess the frequency of "take" (defined as the development of an erythematous papule, vesicle, and/or eschar with or without underlying induration) following vaccination with either the DVC-LVS or USAMRIID-LVS vaccine; and (Immunogenicity): assess the rate of seroconversion following vaccination with either the DVC-LVS or the USAMRIID-LVS vaccine as measured by a tularemia-specific microagglutination assay. The secondary objectives are: (Safety): assess the incidence of adverse events (AEs) following vaccination with either the DVC-LVS or the USAMRIID-LVS vaccine; (Take): assess "take" frequency and difference between vaccine groups as assessed by an independent committee following vaccination with either the DVC-LVS or USAMRIID- LVS vaccine; and (Immunogenicity): assess antibody responses for each group following vaccination with DVC-LVS or USAMRIID-LVS vaccine as measured by a tularemia-specific microagglutination assay. Parent protocol to sub-study 10-0019.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females between the ages of 18 and 45 years, at the day of vaccination
* If the subject is female and of childbearing potential, negative serum pregnancy test at screening and negative urine or serum pregnancy test within 24 hours prior to vaccination.
* If the subject is female and of childbearing potential, she agrees to practice abstinence from sexual intercourse with men (vaginal penetration by a penis, coitus) or use acceptable contraception, for 56 days following vaccination in order to avoid pregnancy:

  1. A woman is considered of childbearing potential unless post-menopausal (greater than or equal to 1 year without menses) or surgically sterilized (tubal ligation, bilateral oophorectomy, or hysterectomy)
  2. Acceptable contraception methods are restricted to effective devices [intrauterine devices (IUDs), NuvaRing®] or licensed hormonal products with use of method for a minimum of 30 days prior to vaccination, condoms with spermicidal agents, monogamous relationship with a vasectomized partner or successful Essure placement with documented confirmation test at least 3 months after the procedure.
* All clinical laboratory values must be within normal limits for age and gender with the following exceptions:

  * White Blood Cell Count: 3.0-10.8 thou/mcl.
  * Absolute Neutrophil count: >/= 1.5 thou/mcl
  * ALT, AST and LDH </= 1.25 x ULN
  * Glucose: </= 115 mg/dl
  * Creatinine: values lower than the normal range are not exclusionary
* Completion of Volunteer Questionnaire
* Willingness to comply with protocol requirements
* Provides informed consent before any protocol procedures are performed
* Availability for follow up for 6 months after vaccination

Exclusion Criteria:

* Current use of antibiotics or antibiotic treatment within last 7 days.
* Current treatment with chemotherapy.
* Use of immunosuppressive or immunomodulatory agents including parenteral, inhaled, or oral corticosteroids within the last 4-weeks. Use of corticosteroid nasal sprays is permissible. Persons who have used topical steroid can be enrolled after their therapy is completed.
* History of splenectomy.
* Has been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years. ((Subjects with a psychiatric disorder (not meeting exclusion criteria, e.g. attention-deficit hyperactivity disorder) that is controlled for a minimum of 3 months and the investigator has determined that the subject's mental status will not compromise the subject's ability to comply with protocol requirements may be enrolled)).
* The subject is taking any of the following psychiatric drugs:

aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate.

* The subject is taking more than one antidepressant drug not included in the list above ((Subjects taking only one antidepressant drug (not listed in excluded psychiatric drugs) who are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study provided the investigator determines the subjects' mental status will not compromise the subjects' ability to comply with protocol requirements.
* History of receiving blood or blood products (such as blood transfusion, platelet transfusion, immunoglobulins, hyperimmune serum) in the previous three months.
* Receipt of licensed inactivated vaccine 14 days prior to vaccination or planned receipt of licensed inactivated vaccine within 14 days post vaccination.
* Receipt of licensed live attenuated vaccine within 30 days prior to vaccination or planned receipt of licensed live attenuated vaccine within 28 days post vaccination.
* Use of any other experimental agent within 30 days prior to vaccination and for the duration of the study.
* Previous vaccination against tularemia.
* Previous treatment for tularemia or history of exposure to tularin.
* Known hypersensitivity to gelatin or other components contained in the vaccine (e.g. glucose cysteine hemin agar).
* History of sensitivity to streptomycin or tetracyclines (including doxycycline).
* History of a chronic medical conditions including, but not limited to, disorders of the liver, kidney, lung, heart or nervous system, or other metabolic and autoimmune/inflammatory conditions that would either interfere with the accurate assessment of the safety, "take" or immunogenicity objectives.
* Presence of an acute condition, including, but not limited to, disorders of the liver, kidney, lung, heart, nervous system, or metabolic and autoimmune inflammatory condition that would interfere with the accurate assessment of the safety, "take" and immunogenicity objectives.
* History of anaphylaxis or serious adverse events following immunization.
* History of alcohol or drug abuse in the past five years or current abuse of alcohol or drugs that in the opinion of the Investigator may interfere with the subject's ability to comply with trial procedures.
* Women that are lactating.
* Acute illness including temperature >100.4 degrees Fahrenheit within one week of vaccination.
* Positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B surface antibody (HBsAg).
* Household contact with infants (children < 1 year), pregnant women, or immunosuppressed individuals, or occupation involving significant contact (e.g., HIV clinic nurse) with infants (children < 1 year), pregnant women, or immunosuppressed individuals, expected to occur in the 14 days after vaccination.
* Identification of any condition that, in the opinion of the investigator, would jeopardize the safety of the subject following vaccination.
* Significant dermatologic disorder (such as eczema, psoriasis). Significant dermatologic disorder includes a history of keloid formation.
* Tattoo(s) in the area of the vaccination sites or evidence of prior injury or damage of the skin at the vaccination sites (e.g. scarring subsequent to burn).
* The presence of any prosthetic implant (such as joint, ventriculoperitoneal shunt, cardiac valve).
* History of malignancy, including hematologic, melanoma skin cancer. Subjects with squamous cell or basal cell carcinoma are eligible provided the areas affected are not in close proximity to the vaccination sites and any sites that were resected are well healed.
* Donation of a unit of blood within 56 days prior to vaccination and/or planned blood donation within 56 days after vaccination (prior to Visit 8).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety: incidence of vaccine-associated serious adverse events (SAEs). | Throughout the course of the study.
Immunogenicity: proportion of subjects that seroconvert (greater than or equal to 4-fold rise in antibody titer) as measured by a tularemia-specific microagglutination assay. | Visits 7 or 8 post vaccination (Day 28 or Day 56).
Safety: incidence of Grade 3 or 4 laboratory values. | Through Day 28 of the study.
Proportion of subjects that develop a positive "take" response, as assessed by the clinical site, defined as the development of an erythematous papule, vesicle, and/or eschar with or without underlying induration. | By study Visit 5 (7-9 days post vaccination).

SECONDARY OUTCOMES:
Take: proportion of subjects that develop a positive "take" response, as assessed by an independent blinded "take committee," following review of photographs taken of the vaccination and placebo sites. | Study Visit 5 (7-9 days post vaccination).
Safety: occurrence of solicited systemic AEs. | Within 28 days post vaccination.
Take: difference in the proportion of subjects that develop a positive "take" response between the two vaccine groups as assessed by an independent blinded "take committee". | Study Visit 5 (7-9 days post vaccination).
Safety: occurrence of solicited local adverse events (AE)s. | Within 28 days post vaccination.
Immunogenicity: geometric mean titers (GMT) of peak microagglutination titer for each arm of the study. For each subject, the peak titer is defined by the maximum titer among all the available measures. | Visits 6, 7 and 8 post vaccination (Day 14, Day 28 and Day 56)..
Take: difference in the proportion of subjects that develop a positive "take" response between the two vaccine groups as assessed by the clinical site. | Study Visit 5 (7-9 days post vaccination).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - University of Iowa - Vaccine Research & Education Unit, Iowa City, Iowa
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas

REFERENCES:
- [Derived] Goll JB, Bosinger SE, Jensen TL, Walum H, Grimes T, Tharp GK, Natrajan MS, Blazevic A, Head RD, Gelber CE, Steenbergen KJ, Patel NB, Sanz P, Rouphael NG, Anderson EJ, Mulligan MJ, Hoft DF. The Vacc-SeqQC project: Benchmarking RNA-Seq for clinical vaccine studies. Front Immunol. 2023 Jan 19;13:1093242. doi: 10.3389/fimmu.2022.1093242. eCollection 2022. PMID 36741404
- [Derived] Mulligan MJ, Stapleton JT, Keitel WA, Frey SE, Chen WH, Rouphael N, Edupuganti S, Beck A, Winokur PL, El Sahly HM, Patel SM, Atmar RL, Graham I, Anderson E, El-Kamary SS, Pasetti MF, Sztein MB, Hill H, Goll JB; DMID 08-0006 Tularemia Vaccine Study Group. Tularemia vaccine: Safety, reactogenicity, "Take" skin reactions, and antibody responses following vaccination with a new lot of the Francisella tularensis live vaccine strain - A phase 2 randomized clinical Trial. Vaccine. 2017 Aug 24;35(36):4730-4737. doi: 10.1016/j.vaccine.2017.07.024. Epub 2017 Jul 24. PMID 28750854